CLINICAL TRIAL: NCT05587712
Title: A Phase 2 Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Sotatercept (MK-7962) in Children From 1 to Less Than 18 Years of Age With PAH on Standard of Care
Brief Title: Study to Evaluate Sotatercept (MK-7962) in Children With Pulmonary Arterial Hypertension (PAH) (MK-7962-008)
Acronym: MOONBEAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7962-008; MK-7962-008 (Other: MSD); 2023-504861-22-00 (Registry Identifier: EU CT); U1111-1290-2858 (Registry Identifier: UTN); 2022-000478-25 (EudraCT Number)
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Children ≥1 to <18 years old (Experimental): Participants will receive a subcutaneous (SC) injection every 3 weeks (Q3W) of 0.3 mg/kg. Dosage may be adjusted based on protocol-specific guidelines.
  Interventions: Drug: Sotatercept

INTERVENTIONS:
Drug: Sotatercept — SC injection every 3 weeks (Q3W) of 0.3 mg/kg. Dosage may be adjusted based on protocol-specific guidelines.
  Other Names: MK-7962

SUMMARY:
The primary objectives of the study are to evaluate the safety and tolerability, and pharmacokinetics (PK) of sotatercept over 24 weeks of treatment in children ≥1 to <18 years of age with PAH World Health Organization (WHO) Group 1 on standard of care (SoC). There is no formal hypothesis.

ELIGIBILITY:
Inclusion Criteria

* Documented, historic diagnostic right heart catheterization (RHC) any time before Screening confirming the diagnosis of PAH WHO Group 1 in any of the following subtypes:
* Idiopathic pulmonary arterial hypertension (IPAH)
* Heritable PAH
* Drug/toxin-induced PAH
* PAH associated with connective tissue disease
* PAH-congenital heart disease (CHD) with shunt closure >6 months before Screening and subsequently confirmed by RHC before Screening
* PAH with coincidental shunt.
* Must be on a stable dose(s) of background PAH therapy (phosphdiesterase-5 (PDE5) inhibitors, endothelin receptor antagonists (ERAs), soluble guanylate cyclase stimulators (sGCS), or prostanoids [including subcutaneous and intravenous])
* If male, agree to the following during the intervention period and for at least 16 weeks (112 days) after the last dose of study intervention:
* Abstains from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agrees to remain abstinent or
* Uses contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause, documented from the site personnel's review of the participant's medical records, medical examination, or medical history interview) as detailed below:
* Uses a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.
* If female, must be either not a WOCBP or use a contraceptive method that is highly effective or be abstinent from heterosexual intercourse during the intervention period and for at least 16 weeks (112 days) after the last dose of study intervention
* If male, agrees to refrain from donating blood or sperm for the duration of the study and for 16 weeks (112 days) after the last dose of study intervention
* If female, agrees to refrain from donating blood, eggs, or ovum for the duration of the study and for at least 16 weeks (112 days) after the last dose of study intervention

Exclusion Criteria

* History of left-sided heart disease, including valvular disease (eg, moderate or greater mitral or aortic regurgitation or stenosis), left ventricular outflow tract obstruction, and/or left heart failure (eg, restrictive or dilated cardiomyopathy)
* Severe (as based on the opinion of the investigator) congenital or developmental abnormalities of the lung, thorax, and/or diaphragm
* History of Eisenmenger syndrome, Potts shunt, or atrial septostomy
* Unrepaired or residual cardiac shunt
* Diagnosis of pulmonary veno-occlusive diseases, pulmonary capillary hemangiomatosis, or overt signs of capillary and/or venous involvement
* PAH associated with portal hypertension
* Known visceral (lung, liver, or brain) arteriovenous malformation(s)
* History of full or partial pneumonectomy
* Untreated more than mild obstructive sleep apnea
* History of known pericardial constriction
* Family history of sudden cardiac death or long QT syndrome
* Any current or prior history of symptomatic coronary disease (myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery, or cardiac anginal chest pain) within 6 months before Screening
* Cerebrovascular accident within 3 months before Screening
* Prior exposure to sotatercept or luspatercept or has had an allergic reaction to any of their excipients

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2028-09-21 (Estimated); Study Completion 2028-09-21 (Estimated)

PRIMARY OUTCOMES:
Serum Trough Concentration (Ctrough) of Sotatercept | Predose Day 1, Day 21, Day 42, Day 63, Day 84, Day105, Day 126, Day 147, Day 168, Day 189. Postdose Day 7, Day 14, Day 64, Day 69 and Day 76
  Ctrough was the lowest concentration of Sotatercept in serum just before the next dose. Blood samples will be collected at multiple time points to estimate the Ctrough of Sotatercept.
Area Under the Curve at Steady State (AUCss) of Sotatercept | Predose Day 1, Day 21, Day 42, Day 63, Day 84, Day105, Day 126, Day 147, Day 168, Day 189. Postdose Day 7, Day 14, Day 64, Day 69 and Day 76
  Blood samples will be collected at multiple time points to estimate the AUCss of Sotatercept.
Area Under the Curve from 0 to 3 weeks (AUC0-3 weeks) of Sotatercept | Predose Day 1, Day 7, Day 14, and Predose Day 21
  Blood samples will be collected at Predose Day 1, Day 7, Day 14, and Predose Day 21 to estimate the AUC0-3 weeks of Sotatercept.
Percentage of Participants Who Experience at Least 1 Adverse Event (AE) | Up to 24 weeks
  An AE is any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The percentage of participants with 1 or more AEs will be assessed.
Percentage of Participants Who Discontinue Study Drug Due to an AE | Up to 24 weeks
  An AE is any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. The percentage of participants who discontinued the study drug due to an AE regardless of study completion status will be assessed.
Laboratory Parameter (Hematology): Concentration of Hemoglobin | Up to 24 weeks
  Hematological parameters will be investigated in blood samples from participants by means of clinical laboratory assays and evaluated by the investigator. The concentration of hemoglobin will be presented.
Laboratory Parameter (Hematology): Hematocrit | Up to 24 weeks
  Hematological parameters will be investigated in blood samples from participants by means of clinical laboratory assays and evaluated by the investigator. The hematocrit will be presented.
Laboratory Parameter (Hematology): Red Blood Cell (RBC) Count | Up to 24 weeks
  Hematological parameters will be investigated in blood samples from participants by means of clinical laboratory assays and evaluated by the investigator. The RBC count will be presented.
Laboratory Parameter (Hematology): Reticulocyte Count | Up to 24 weeks
  Hematological parameters will be investigated in blood samples from participants by means of clinical laboratory assays and evaluated by the investigator. The reticulocyte count will be presented.
Laboratory Parameter (Hematology): Platelet Count | Up to 24 weeks
  Hematological parameters will be investigated in blood samples from participants by means of clinical laboratory assays and evaluated by the investigator. The platelet count will be presented.
Blood Pressure (BP) | Up to 24 weeks
  BP will be assessed while the participant was seated after a period of rest in a quiet setting with no distractions (eg, television and cell phones).
Titer of Anti-drug Antibody (ADA) to Sotatercept | Up to 24 weeks
  ADA to Sotatercept will be assessed.

SECONDARY OUTCOMES:
Mean Change from Baseline in 6-Minute Walk Distance (6MWD) (Cohorts 1 and 2) | Baseline and Week 24
  6MWD will be assessed using the 6-minute walk test (6MWT).
Mean Change from Baseline in Tricuspid Annular Plane Systolic Excursion (TAPSE) | Baseline and Week 24
  A two-dimensional echocardiogram (ECHO) will be performed with the results interpreted by a blinded independent central review (BICR) at baseline and after 24 weeks of treatment. The change from baseline in TAPSE will be reported.
Mean Change from Baseline in Pulmonary Artery Systolic Pressure (PASP) | Baseline and Week 24
  A two-dimensional ECHO will be performed with the results interpreted by a BICR at baseline and after 24 weeks of treatment. The change from baseline in PASP will be reported.
Mean Change from Baseline in Right Ventricular Fractional Area Change (RVFAC) | Baseline and Week 24
  A two-dimensional ECHO will be performed with the results interpreted by a BICR at baseline and after 24 weeks of treatment. The change from baseline in RVFAC will be reported.
Mean Change from Baseline in Eccentricity Index | Baseline and Week 24
  A two-dimensional ECHO will be performed with the results interpreted by a BICR at baseline and after 24 weeks of treatment. The change from baseline in eccentricity index will be reported.
Mean Change from Baseline in Right Ventricular (RV) Function (Cohorts 1 and 2) | Baseline and Week 24
  Cardiac magnetic imaging (MRI) will be performed with the results interpreted by a BICR at baseline and after 24 weeks of treatment. The change from baseline in eccentricity index will be reported.
Mean Change from Baseline on Cardiac Output (Cohorts 1 and 2) | Baseline and Week 24
  Cardiac magnetic imaging (MRI) will be performed with the results interpreted by a BICR at baseline and after 24 weeks of treatment. The change from baseline in cardiac output will be reported.
Mean Change from Baseline in Pulmonary Arterial Pressure (PAP) (Cohorts 1 and 2) | Baseline and Week 24
  Cardiac magnetic imaging (MRI) will be performed with the results interpreted by a BICR at baseline and after 24 weeks of treatment. The change from baseline in PAP will be reported.
Mean Change from Baseline in Pediatric Quality of Life (PedsQL) Generic Score | Baseline and Week 24
  PedsQL Measurement Model is a modular approach to measuring health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. The change from baseline in the PedsQL generic core scale will be reported.
Mean Change from Baseline in N-terminal Prohormone B-type Natriuretic Peptide (NT-proBNP) | Baseline and Week 24
  The change from baseline in plasma NT-proBNP levels will be reported.
Percentage of Participants Who Either Improved or Maintained Their World Health Organization Functional Class (WHO FC) | Baseline and Week 24
  The severity of an individual's PAH symptoms will be graded using the WHO FC system. WHO functional classification for PAH range from Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity) and Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest). The change from baseline in WHO FC will be classified into "Improved", "No change" and "Worsened". Improvement = reduction in FC, worsened = increase in FC and no change = no change in FC.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (35):
- United States (10):
  - The Regents of the University of California - Los Angeles (UCLA Pediatrics) ( Site 1606), Los Angeles, California
  - Stanford University School of Medicine ( Site 1603), Palo Alto, California
  - UCSF Benioff Children's Hospital San Francisco ( Site 1611), San Francisco, California
  - Children's Hospital Colorado ( Site 1609), Aurora, Colorado
  - Children's National Medical Center ( Site 1600), Washington D.C., District of Columbia
  - Cincinnati Children's Hospital Medical Center ( Site 1602), Cincinnati, Ohio
  - Children's Hospital of Philadelphia (CHOP) ( Site 1608), Philadelphia, Pennsylvania
  - Monroe Carell Jr. Children's Hospital ( Site 1601), Nashville, Tennessee
  - Seattle Children's Hospital ( Site 1605), Seattle, Washington
  - Children's Wisconsin ( Site 1610), Milwaukee, Wisconsin
- The Children's Hospital at Westmead ( Site 0001), Westmead, New South Wales, Australia
- Colombia (3):
  - Clinica Somer-Unidad de Investigacion y Docencia ( Site 0205), Rionegro, Antioquia
  - Fundación Valle del Lili ( Site 0200), Cali, Valle del Cauca Department
  - Clínica Imbanaco S.A.S ( Site 0203), Cali, Valle del Cauca Department
- France (3):
  - CHU de Toulouse - Hôpital des Enfants ( Site 0302), Toulouse, Haute-Garonne
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone ( Site 0303), Marseille, Provence-Alpes-Côte d'Azur Region
  - Hôpital Universitaire Necker Enfants Malades ( Site 0300), Paris
- Germany (3):
  - Universitaetsklinikum Heidelberg ( Site 0401), Heidelberg, Baden-Wurttemberg
  - Klinikum der Universität München Großhadern ( Site 0404), München, Bavaria
  - Medizinische Hochschule Hannover ( Site 0405), Hanover, Lower Saxony
- Israel (2):
  - Schneider Children's Medical Center ( Site 0603), Petah Tikva
  - Sheba Medical Center ( Site 0601), Ramat Gan
- University Medical Center Groningen ( Site 0900), Groningen, Netherlands
- Poland (2):
  - Centrum Zdrowia Dziecka w Warszawie-Klinika Kardiologii ( Site 1103), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Kardiologii Dziecięcej i Wad Wrodzonych Serca ( Site 1102), Gdansk, Pomeranian Voivodeship
- Wits Clinical Research-Wits Clinical Research Bara ( Site 1201), Johannesburg, Soweto, Gauteng, South Africa
- Spain (4):
  - Hospital Universitario Ramón y Cajal ( Site 1300), Madrid, Madrid, Comunidad de
  - Hospital Universitari i Politecnic La Fe ( Site 1303), Valencia, Valencia
  - Hospital Universitari Vall d'Hebron ( Site 1302), Barcelona
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON ( Site 1301), Madrid
- Turkey (Türkiye) (4):
  - Hacettepe Universite Hastaneleri ( Site 1400), Ankara
  - Gazi University Health Research and Application Center Gazi -Çocuk Sağlığı ve Hastalıkları Anabilim ( Site 1402), Ankara
  - Ankara Bilkent Şehir Hastanesi. ( Site 1403), Ankara
  - Mehmet Akif Ersoy Research and Training Hospital ( Site 1404), Istanbul
- Great Ormond Street Hospital For Children NHS Foundation Trust ( Site 1500), London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26279&tenant=MT_MSD_9011